Impact of Retro-molar pad carving on complete denture wearers satisfaction and quality of life: a cross-over, double-blind clinical trial.

| Statistics | 27/8/2025 |
|---|---|
| Samiha Sartawi <sup>a*</sup> ,, , | , Mahmoud K. AL-Omiri <sup>z</sup> |
| <sup>a</sup> Department of Fixed and Removable Prostho<br>Jordan, Amman 11942, Jordan. Email: | odontics, School of Dentistry, The University of |
| <sup>z</sup> Department of Fixed and Removable Prostho<br>Jordan, Amman 11942, Jordan. Email: <u>alomir</u> i | odontics, School of Dentistry, The University of im@yahoo.co.uk |
| Corresponding author: | |
| Dr Samiha Sartawi | |
| Department of Fixed and Removable Prosthod | lontics, School of Dentistry, |
| The University of Jordan, Queen Rania Street, | |
| Amman 11942, Jordan | |
| Email: | |

## **Statistical analysis:**

The SPSS computer software (IBM SPSS Statistics v21.0; IBM Corp., USA) was utilized for the statistical analysis of the collected data in this study. The significance of the conducted statistical results was considered at two tailed  $\alpha$  of .05. Normal distribution of the data was tested utilizing the Shapiro-Wilk test and the skewness test considering skewness z-score threshold values range from -3.29 to +3.29. All the continuous variables were not normally distributed, except for age and OHIP scores before treatment. Descriptive statistics for normally distributed continuous variables (age and OHIP scores before treatment) included the mean, standard error, standard deviation, median, maximum value, minimum value, and confidence intervals. Meanwhile, descriptive statistics for the non-normally distributed continuous variables included the mean, standard deviation, median, interquartile range, minimum value, and maximum value. Categorical variables in this study (presence of redness, erosion, keratosis, ulceration, and denture fissuratum) were presented as frequencies and percentages.

The Wilcoxon Signed Ranks test was used to test paired differences in satisfaction ratings, dentist's evaluations, and OHIP-EDENT scores after using carved and non-carved lower dentures. The Mann Whitney U test was utilized to identify differences in satisfaction ratings, dentist's evaluations, and OHIP-EDENT scores between genders. Spearman's Rho rank correlations were used to identify the correlations between satisfaction ratings, dentist's evaluations, and OHIP-EDENT scores. Associations between identification of lesions following denture use (presence of redness, erosion, keratosis, ulceration, and denture fissuratum) and having the retromolar pad area of the lower denture carved or not were tested via Fisher's Exact test.

The multiple linear regression analysis was used to identify the contribution of having the retromolar pad area carved or not, satisfaction ratings, and dentist evaluation towards the prediction of OHIP-EDENT scores considering the confounding effects of gender and age.

The calculated sample size was 46 participants. A priori power analysis based on linear multiple regression test (G\*Power, version 3.1.9.7; Heinrich-Heine University) calculated the minimum sample size to be 46 participants. The calculation considered a significance level ( $\alpha$ ) of .05, a statistic power (1 –  $\beta$ ) of 0.8, and an effect size of 0.3. Extra participants were recruited to balance for participant drop outs and secure the required minimum sample size. Fifty participants were recruited for the study, and none of participants was lost during the investigation (drop out ratio was 0%). Therefore, 50 participants were finally recruited and completed the study, and had their data collected and analyzed.

## Results

The data was collected from a total of 49 participants (23 females and 27 males), and was then processed and analyzed. Participants age ranged from 40 to 78 years old (mean age= 62.8 years old, SD= 8.01, SE= 1.145, median= 63.0, 95% CI= 60.51 - 65.12).

Table 1 demonstrates the descriptive statistics for continuous variables in this study including dentist evaluations of dentures, patients' satisfaction with dentures, and OHIP-EDENT scores among the participants of this study. Paired comparisons of carved and non-carved lower dentures showed that patient satisfaction with retention at function (P=.002) and comfort during the use of carved lower dentures (P=.026) were significantly higher than non-carved lower dentures (Table 1). Furthermore, the patients demonstrated a tendency to be more satisfied with denture retention at rest as well as during eating when used carved lower dentures in comparison to non-carved ones. This difference was not significant but was close to be significant (P=.052,

Table 1). In addition, carved lower dentures were associated with lower OHIP scores (better impacts on oral health) than the non-carved lower dentures; however, the difference was not significant (P= .055, Table 1). Nevertheless, this tendency was confirmed by the Mann Whitney U test as a significant difference was found in the OHIP scores between carved and non-carved lower dentures (MWU= 887.0, Z= -2.241, P= .025). The carved lower dentures were associated with lower OHIP scores indicating better impacts on oral health than the non-carved dentures.

Table 2 presents the distribution (frequencies and percentages) of redness, erosion, keratosis, ulceration, and denture fissuratum following the use of the tested complete denture designs during this study. Redness was the most observed mucosal change, 18.4% with non-carved dentures and 12.2% with carved dentures. No significant differences in mucosal changes were observed between carved and non-carved lower dentures (P> .05, Table 2).

The results showed that the dentists assigned better ratings for upper dentures in comparison to non-carved lower dentures regarding to denture retention (P=.004) as well as denture support (P=.011) (Table 3). In addition, patients assigned significantly lower pain scores for upper dentures than non-carved lower dentures (P=.008, Table 3). Also, patients reported higher satisfaction with upper dentures considering denture retention at rest (P=.035), denture retention at function (P<.001), and comfort during denture use (P<.001) in comparison to non-carved lower dentures (Table 3). In contrast, no significant differences between upper dentures and lower carved dentures regarding any dentist ratings or patient satisfaction for any evaluated factor (P>.05 Table 3).

Gender base variations showed that females were assigned higher dentist ratings for retention of non-carved lower dentures (P= .031), stability of lower non-carved dentures (P= .003), support of lower non-carved dentures (P= .014), esthetics of lower carved (P= .007) and

non-carved dentures (P=.001), stability of upper denture (P=.035), and esthetics of upper denture (P=.004) (Table 4). Also, females reported more pain with lower carved dentures in comparison to males (P=.015, Table 4). In addition, females assigned higher satisfaction ratings regarding retention during function of lower non-carved denture (P=.015), comfort of lower non-carved denture (P=.007), retention at rest for upper denture (P=.007), retention at function for upper denture (P=.002), comfort of upper denture (P=.001), and retention during eating with upper denture and lower non-carved denture (P=.045) (Table 4).

Table 5 presents correlations between age, patient satisfaction, and OHIP scores. The results shows that older patients were more comfortable with upper dentures than younger patients (Spearman Rho= 0.309, P= .031, Table 5). Also, higher pain scores were associated with higher OHIP scores (i.e. worse impacts) after using carved (P= .001) and non-carved (P< .001) lower dentures (Table 5). In addition, lower OHIP scores (i.e. better impacts) were associated with higher satisfaction with retention at rest, retention at function, denture comfort, general satisfaction with dentures, retention during eating, and retention during speaking after using carved or non-carved lower dentures (P< .05, Table 5). Besides, correlations between age and dentist rating of dentures showed that older participants were found to have better dentist ratings of retention (Sperman Rho= 0.402, P= .004) and higher stability (Spearman Rho= 0.402, P= .003) of upper dentures than younger participants.

A multiple linear regression analysis was used to identify the contribution of having the retromolar pad area carved or not, satisfaction ratings, and dentist evaluation of dentures towards the prediction of OHIP scores considering the confounding effects of gender and age (Table 6). Being a female, having lower dentist ratings of denture esthetics, and having more pain due to lower dentures were associated with higher scores of OHIP indicating worse oral health impacts

of the prosthesis (P<.05, Table 6). Being a female was associated with an increase of OHIP scores by 4 units (P=.007). Also, for each decreased unit of dentist ratings of denture esthetics, the OHIP scores were increased by 2 units (P=.018). Furthermore, for each increased unit of pain levels due to lower dentures, the OHIP scores were increased by 0.7 units (P=.020) (Table 6).

Further multiple linear regression analyses were conducted to identify the contribution of having the retromolar pad area carved or not and dentist evaluation of dentures towards the prediction of patient satisfaction with different denture aspects considering the confounding effects of gender and age (Table 7). The results showed that carved lower dentures were associated with 1.144 times higher satisfaction with lower denture retention during function (P= .040, Table 7). Dr Samiha please note that Being carved or not was significant predictor for retention of the denture during function. Besides, patients satisfaction with lower denture retention at rest was decreased by 0.053 unit for each year increase in the age (P= .027, Table 7). Also, being a female was associated with higher patient satisfaction with lower denture retention at rest (B= 0.970, P= .033), lower denture retention at function (B= 1.404, P= .027), lower denture comfort (B= 1.374, P= .007), general satisfaction with upper and lower dentures (B= 1.361, P= .002), and retention of upper and lower dentures during eating (B= 0.978, P= .036) (Table 7).

In addition, higher levels of perceived pain due to lower dentures were associated with lower levels of satisfaction with lower denture retention at rest (B=-0.184, P=.032), lower denture retention at function (B=-0.365, P=.002), lower denture comfort (B=-0.440, P<.001), general satisfaction with upper and lower dentures (B=-0.254, P=.002), retention of upper and lower dentures during eating (B=-0.320, P<.001), and retention of upper and lower dentures during

speaking (B= -0.235, P= .005) (Table 7). Furthermore, higher dentist ratings of lower denture stability (Dr Samiha please note for the discussion that this could be explained by that stability is related to each of retention, support and occlusion) was associated with higher patient satisfaction with lower denture retention at rest (B= 0.527, P= .037), lower denture retention at function (B= 0.958, P= .005), and lower denture comfort (B= 0.723, P= .011) (Table 7).

## **Tables**

**Table 1.** Descriptive statistics for continuous variables including dentist evaluations of dentures, patients' satisfaction with dentures, and OHIP-EDENT scores among the participants of this study (N=50).

| | | | | | | | Paired com | parisons |
|---|---|---|---|---|---|---|---|---|
| | Descri | iptive st | atistic | S | | | of NCLD a | and CLD |
| Variable | Mean | SD | Med | Min | Max | IQR | Z | P |
| Dentist evaluation of dentures | | | | | | | | |
| Retention of NCLD | 8.02 | 1.882 | 8.5 | 2.0 | 10.0 | 2.8 | -1.357 | .175 |
| Retention of CLD | 8.34 | 2.011 | 8.5 | 2.0 | 10.0 | 1.8 | | |
| Stability of NCLD | 8.36 | 1.454 | 8.5 | 2.0 | 10.0 | 1.5 | -1.906 | .057 |
| Stability of CLD | 8.63 | 1.642 | 9.0 | 1.0 | 10.0 | 1.0 | | |
| Support of NCLD | 8.78 | 1.295 | 9.0 | 2.0 | 10.0 | 1.0 | -1.053 | .292 |
| Support of CLD | 9.05 | 0.694 | 9.0 | 7.0 | 10.0 | 1.0 | | |
| Esthetic of NCLD | 8.87 | 0.846 | 9.0 | 6.5 | 10.0 | 1.0 | 223 | .824 |
| Esthetic of CLD | 8.90 | 0.878 | 9.0 | 6.0 | 10.0 | 1.0 | | |
| Retention of upper denture | 8.89 | 1.217 | 9.0 | 5.5 | 10.0 | 1.5 | | |
| Stability of upper denture | 8.66 | 1.192 | 8.5 | 4.5 | 10.0 | 1.5 | | |
| Support of upper denture | 9.21 | 0.707 | 9.5 | 7.0 | 10.0 | 1.3 | | |
| Esthetic of upper denture | 8.90 | 0.835 | 9.0 | 7.0 | 10.0 | 1.0 | | |
| Patient satisfaction with dentures | | | | | | | | |
| Pain due to NCLD | 2.08 | 2.745 | 0.0 | 0.0 | 10.0 | 4.0 | -1.901 | .057 |
| Pain due to CLD | 1.20 | 2.336 | 0.0 | 0.0 | 8.0 | 1.0 | | |
| Retention at rest of NCLD | 8.06 | 2.313 | 9.0 | 2.0 | 10.0 | 3.0 | -1.943 | .052 |
| Retention at rest of CLD | 8.67 | 2.025 | 9.0 | 0.0 | 10.0 | 2.0 | | |
| Retention at function of NCLD | 6.33 | 3.085 | 7.0 | 0.0 | 10.0 | 5.0 | -3.054 | .002 |
| Retention at function of CLD | 7.59 | 2.684 | 8.0 | 0.0 | 10.0 | 3.5 | | |
| Comfort of NCLD | 7.18 | 2.796 | 8.0 | 0.0 | 10.0 | 4.0 | -2.225 | .026 |
| Comfort of CLD | 8.00 | 2.415 | 9.0 | 0.0 | 10.0 | 3.0 | | |
| Insertion of NCLD | 9.92 | 1.891 | 10.0 | 2.0 | 20.0 | 0 | 071 | .943 |
| Insertion of CLD | 9.84 | 0.514 | 10.0 | 8.0 | 11.0 | 0 | | |
| Pain due to upper denture | 0.67 | 2.115 | 0.0 | 0.0 | 10.0 | 0 | | |
| Retention at rest for upper denture | 8.84 | 1.724 | 9.0 | 2.0 | 10.0 | 1.0 | | |
| Retention at function for upper denture | 8.41 | 1.848 | 9.0 | 3.0 | 10.0 | 3.0 | | |
| Comfort for upper denture | 8.74 | 1.765 | 9.0 | 2.0 | 10.0 | 2.0 | | |
| Insertion for upper denture | 9.80 | 0.456 | 10.0 | 8.0 | 10.0 | 0 | | |
| General satisfaction with upper and | 7.88 | 2.304 | 9.0 | 0.0 | 10.0 | 2.8 | 980 | .327 |
| non carved lower dentures | | | | | | | | |
| General satisfaction with upper and | 8.37 | 1.551 | 9.0 | 4.0 | 10.0 | 2.0 | | |
| carved lower dentures | | | | | | | | |
| Retention during eating with upper and | 7.25 | 2.260 | 8.0 | 1.0 | 10.0 | 3.0 | -1.944 | .052 |
| non carved lower dentures | | | | _ | | | | |
| Retention during eating with upper and | 7.98 | 1.953 | 8.0 | 0.0 | 10.0 | 2.5 | | |

| carved lower dentures | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Smile and appearance of upper and | 9.61 | 0.885 | 10.0 | 6.0 | 10.0 | 0.5 | 283 | .777 |
| non carved lower dentures | | | | | | | | |
| Smile and appearance of upper and | 9.65 | 0.694 | 10.0 | 7.0 | 10.0 | 0.5 | | |
| carved lower dentures | | | | | | | | |
| Retention during speaking with upper | 9.14 | 1.414 | 10.0 | 3.0 | 10.0 | 1.0 | 662 | .508 |
| and non carved lower dentures | | | | | | | | |
| Retention during speaking with upper | 9.10 | 2.400 | 10.0 | 0.0 | 20.0 | 2.0 | | |
| and carved lower dentures | | | | | | | | |
| OHIP scores | | | | | | | | |
| OHIP scores before dentures | 22.59 | 10.82 | 20.0 | 4.0 | 48.0 | 17.0 | | |
| OHIP scores after using NCLD | 11.12 | 7.793 | 9.0 | 2.0 | 39.0 | 8.0 | -1.916 | .055 |
| OHIP scores after using CLD | 8.45 | 6.433 | 6.0 | 0.0 | 31.0 | 7.5 | | |

NCLD= Non-carved lower denture, CLD= Carved lower denture, OHIP= Oral Health Impact Profile – 14, SD= Standard deviation, Med= Median, Min= Minimum value, Max= Maximum value, IQR= Interquartile range, Z= Z statistic using Wilcoxon signed ranks test, P= Two-tailed probability value.

**Table 2.** Distribution of redness, erosion, keratosis, ulceration, and denture fissuratum following the use of the tested complete denture designs in this study (N=50).

| | Non | -carved | lower | r denture | Carv | ed lowe | er den | ture | Comparison between | |
|---|---|---|---|---|---|---|---|---|---|---|
| | No | | Yes | Yes | | No | | | carved and non-carv | |
| | | | | | | | | dentures | | |
| Variables | Fre | % | Fre | % | Fre | % | Fre | % | Z | P |
| Redness | 40 | 81.6 | 9 | 18.4 | 43 | 87.8 | 6 | 12.2 | -0.837 | .402 |
| Keratosis | 49 | 100.0 | 0 | 0 | 49 | 100.0 | 0 | 0 | 0 | 1.00 |
| Erosion | 48 | 98.0 | 1 | 2.0 | 47 | 95.9 | 2 | 4.1 | -0.583 | .560 |
| Ulceration | 48 | 98.0 | 1 | 2.0 | 49 | 100.0 | 0 | 0 | -1.000 | .317 |
| Denture Fissuratum | 49 | 100.0 | 0 | 0 | 49 | 100.0 | 0 | 0 | 0 | 1.00 |

Fre= Frequency, %= Percentage. Z= Z statistic using Wilcoxon signed ranks test, P= Two-tailed probability value.

Table 3. Paired comparisons of dentist and patient denture ratings between upper complete dentures and each tested design of lower dentures in this study (N=50).

| Compared pairs | Z | P |
|----------------------------------------------------|--------|------|
| Dentist evaluation of dentures | • | · |
| Retention of NCLD versus upper denture | -2.887 | .004 |
| Retention of CLD versus upper denture | -1.506 | .132 |
| Stability of NCLD versus upper denture | -1.343 | .179 |
| Stability of CLD versus upper denture | 854 | .393 |
| Support of NCLD versus upper denture | -2.558 | .011 |
| Support of CLD versus upper denture | -1.165 | .244 |
| Esthetic of NCLD versus upper denture | -0.019 | .985 |
| Esthetic of CLD versus upper denture | -0.153 | .879 |
| Patient satisfaction with dentures | | |
| Pain due to NCLD versus upper denture | -2.653 | .008 |
| Pain due to CLD versus upper denture | -1.178 | .239 |
| Retention at rest of NCLD versus upper denture | -2.104 | .035 |
| Retention at rest of CLD versus upper denture | -0.285 | .775 |
| Retention at function of NCLD versus upper denture | -4.149 | .000 |
| Retention at function of CLD versus upper denture | -1.831 | .067 |
| Comfort of NCLD versus upper denture | -3.546 | .000 |
| Comfort of CLD versus upper denture | -1.700 | .089 |
| Insertion of NCLD versus upper denture | -0.688 | .491 |
| Insertion of CLD versus upper denture | -0.500 | .617 |

NCLD= Non-carved lower denture, CLD= Carved lower denture, Z= Z statistic using Wilcoxon signed ranks test, P= Two-tailed probability value.

Table 4. Gender based differences of dentist ratings of the dentures, patient satisfaction with dentures, and OHIP scores among the study sample (N=50).

| Variable | Male | | Female | | Gender | Gender difference | |
|---|---|---|---|---|---|---|---|
| Variable | Mean | SD | Mean | SD | MWU | Z | P |
| Age | 61.07 | 6.821 | 64.95 | 8.968 | 204.0 | -1.873 | .061 |
| <b>Dentist evaluation of dentures</b> | | | | | | | |
| Retention of NCLD | 7.48 | 2.040 | 8.68 | 1.452 | 191.0 | -2.153 | .031 |
| Retention of CLD | 7.85 | 2.437 | 8.93 | 1.105 | 228.5 | -1.401 | .161 |
| Stability of NCLD | 7.83 | 1.647 | 9.00 | 0.831 | 153.5 | -2.931 | .003 |
| Stability of CLD | 8.33 | 1.896 | 9.00 | 1.205 | 213.0 | -1.721 | .085 |
| Support of NCLD | 8.43 | 1.517 | 9.21 | 0.797 | 176.5 | -2.466 | .014 |
| Support of CLD | 9.02 | 0.628 | 9.09 | 0.781 | 267.5 | 611 | .541 |
| Esthetic of NCLD | 8.56 | 0.738 | 9.25 | 0.827 | 133.5 | -3.370 | .001 |
| Esthetic of CLD | 8.65 | 0.806 | 9.21 | 0.882 | 166.5 | -2.691 | .007 |
| Retention of upper denture | 8.63 | 1.276 | 9.21 | 1.087 | 209.0 | -1.808 | .071 |
| Stability of upper denture | 8.32 | 1.360 | 9.09 | 0.781 | 194.0 | -2.107 | .035 |
| Support of upper denture | 9.17 | 0.785 | 9.27 | 0.612 | 283.5 | 279 | .780 |
| Esthetic of upper denture | 8.63 | 0.715 | 9.23 | 0.869 | 157.5 | -2.861 | .004 |
| Patient satisfaction with dentures | 1 | | | • | • | • | |
| Pain due to NCLD | 2.22 | 3.068 | 1.91 | 2.348 | 290.0 | 151 | .880 |
| Pain due to CLD | 0.70 | 1.918 | 1.82 | 2.684 | 198.5 | -2.428 | .015 |
| Pain due to upper denture | 0.30 | 0.912 | 1.14 | 2.965 | 285.0 | 424 | .672 |
| Retention at rest of NCLD | 7.33 | 2.801 | 8.96 | 0.999 | 207.0 | -1.860 | .063 |
| Retention at rest of CLD | 8.52 | 1.949 | 8.86 | 2.145 | 257.5 | 841 | .400 |
| Retention at function of NCLD | 5.33 | 3.234 | 7.55 | 2.444 | 177.0 | -2.430 | .015 |
| Retention at function of CLD | 7.22 | 2.778 | 8.05 | 2.554 | 231.0 | -1.353 | .176 |
| Comfort of NCLD | 6.22 | 3.017 | 8.36 | 1.989 | 165.5 | -2.682 | .007 |
| Comfort of CLD | 7.82 | 2.419 | 8.23 | 2.448 | 255.0 | 871 | .384 |
| Insertion of NCLD | 9.56 | 1.577 | 10.36 | 2.172 | 266.5 | -1.008 | .313 |
| Insertion of CLD | 9.82 | 0.623 | 9.86 | 0.351 | 294.0 | 094 | .925 |
| Retention at rest for upper denture | 8.26 | 2.087 | 9.55 | 0.671 | 172.0 | -2.687 | .007 |
| Retention at function for upper | 7.67 | 2.019 | 9.32 | 1.086 | 150.5 | -3.074 | .002 |
| denture | | | | | | | |
| Comfort for upper denture | 8.00 | 2.057 | 9.64 | 0.581 | 148.0 | -3.210 | .001 |
| Insertion for upper denture | 9.70 | 0.542 | 9.91 | 0.294 | 246.0 | -1.525 | .127 |
| General satisfaction with upper and | 7.26 | 2.768 | 8.64 | 1.246 | 222.0 | -1.536 | .125 |
| non carved lower dentures | | | | | | | |
| General satisfaction with upper and carved lower dentures | 8.00 | 1.776 | 8.82 | 1.097 | 225.0 | -1.491 | .136 |
| Retention during eating with upper | 6.59 | 2.576 | 8.05 | 1.495 | 198.5 | -2.008 | .045 |
| and non carved lower dentures | 0.39 | 2.370 | 0.03 | 1.473 | 170.3 | -2.008 | .043 |
| Retention during eating with upper and carved lower dentures | 8.07 | 1.639 | 7.86 | 2.316 | 295.0 | 041 | .967 |
| Smile and appearance of upper and | 9.56 | 0.892 | 9.68 | 0.894 | 263.5 | 897 | .370 |

| non carved lower dentures | | | | | | | |
|---|---|---|---|---|---|---|---|
| Smile and appearance of upper and | 9.56 | 0.698 | 9.77 | 0.685 | 240.0 | -1.524 | .127 |
| carved lower dentures | | | | | | | |
| Retention during speaking with upper | 8.96 | 1.698 | 9.36 | 0.954 | 264.0 | 734 | .463 |
| and non carved lower dentures | | | | | | | |
| Retention during speaking with upper | 8.89 | 1.368 | 9.36 | 3.274 | 246.5 | -1.097 | .273 |
| and carved lower dentures | | | | | | | |
| OHIP scores | | | | | | | |
| OHIP scores before dentures | 23.04 | 9.469 | 22.05 | 12.492 | 268.0 | 584 | .559 |
| OHIP scores after using NCLD | 11.07 | 6.644 | 11.18 | 9.174 | 266.5 | 616 | .538 |
| OHIP scores after using CLD | 7.78 | 4.925 | 9.27 | 7.953 | 294.5 | 051 | .959 |

NCLD= Non-carved lower denture, CLD= Carved lower denture, OHIP= Oral Health Impact Profile – 14, SD= Standard deviation, MWU= Mann Whitney U test statistic, Z= Z statistic, P= Two-tailed probability value.

Table 5. Correlations between age, patient satisfaction, and OHIP scores among the study population (N=50).

| Variable | Statistics | Age | OHIP after NCLD | OHIP after CLD |
|---|---|---|---|---|
| Age | Rho | 1.000 | 226 | .047 |
| | P | - | .119 | .746 |
| Pain due to NCLD | Rho | 076 | .554 | .183 |
| | P | .605 | <.001 | .208 |
| Pain due to CLD | Rho | .269 | .205 | .467 |
| | P | .061 | .158 | .001 |
| Pain due to upper denture | Rho | 182 | .166 | 214 |
| | P | .212 | .254 | .139 |
| Retention at rest of NCLD | Rho | 079 | 367 | .017 |
| | P | .591 | .010 | .910 |
| Retention at rest of CLD | Rho | 243 | 175 | 414 |
| | P | .093 | .228 | .003 |
| Retention at function of NCLD | Rho | .162 | 480 | 164 |
| | P | .266 | <.001 | .261 |
| Retention at function of CLD | Rho | 162 | 164 | 511 |
| | P | .267 | .261 | <.001 |
| Comfort of NCLD | Rho | .175 | 518 | 214 |
| | P | .230 | <.001 | .141 |
| Comfort of CLD | Rho | 214 | 223 | 643 |
| | P | .141 | .123 | <.001 |
| Insertion of NCLD | Rho | 012 | 344 | 162 |
| | P | .934 | .016 | .266 |
| Insertion of CLD | Rho | 194 | 365 | 248 |
| | P | .181 | .010 | .086 |
| Retention at rest for upper denture | Rho | .199 | 346 | 192 |
| | P | .170 | .015 | .187 |
| Retention at function for upper | Rho | .229 | 271 | 288 |
| denture | P | .113 | .059 | .045 |
| Comfort for upper denture | Rho | .309 | 339 | 188 |
| | P | .031 | .017 | .196 |
| Insertion for upper denture | Rho | .050 | 341 | 310 |
| | P | .731 | .016 | .030 |
| General satisfaction with upper and | Rho | .041 | 481 | 052 |
| non carved lower dentures | P | .778 | <.001 | .721 |
| General satisfaction with upper and | Rho | .058 | 316 | 491 |
| carved lower dentures | P | .695 | .027 | <.001 |
| Retention during eating with upper | Rho | .260 | 582 | 032 |
| and non carved lower dentures | P | .072 | <.001 | .828 |
| Retention during eating with upper | Rho | 069 | 320 | 459 |
| and carved lower dentures | P | .639 | .025 | .001 |
| Smile and appearance of upper and | Rho | 102 | 290 | 196 |

| non carved lower dentures | P | .484 | .043 | .177 |
|-------------------------------------|-----|------|------|-------|
| Smile and appearance of upper and | Rho | .181 | 359 | 207 |
| carved lower dentures | P | .213 | .011 | .153 |
| Retention during speaking with | Rho | .066 | 435 | 145 |
| upper and non carved lower dentures | P | .655 | .002 | .321 |
| Retention during speaking with | Rho | 016 | 276 | 505 |
| upper and carved lower dentures | P | .911 | .055 | <.001 |
| OHIP score before treatment | Rho | 104 | .253 | 052 |
| | P | .479 | .079 | .722 |

NCLD= Non-carved lower denture, CLD= Carved lower denture, OHIP= Oral Health Impact Profile – 14, Rho= Spearman correlation coefficient, P= Two tailed probability value.

**Table 6.** Linear regression analyses to predict OHIP scores after treatment utilizing the demographic variables, having the lower denture carved or not, dentist ratings of lower dentures, and patient satisfaction with dentures among the study sample (n= 50).

| | | Unst | Co | St Co | | | 95% CI | I for B |
|---|---|---|---|---|---|---|---|---|
| Dependent | | | | | | | Lower | |
| variable | Predictors* | В | SE | Beta | t | P | Bound | Bound |
| OHIP scores | Constant | 63.274 | 13.648 | | 4.636 | <.001 | 36.118 | 90.430 |
| after | Gender | 4.063 | 1.465 | .281 | 2.774 | .007 | 1.149 | 6.977 |
| treatment | Age | 132 | .080 | 146 | -1.645 | .104 | 292 | .028 |
| $R^2 = .468$ | Carved denture or not | -1.324 | 1.222 | 092 | -1.084 | .282 | -3.755 | 1.107 |
| DW=1.837 | Dentist rated lower denture | .314 | .507 | .084 | .619 | .538 | 695 | 1.323 |
| | retention | | | | | | | |
| | Dentist rated lower denture stability | 704 | .793 | 151 | 888 | .377 | -2.282 | .873 |
| | Dentist rated lower denture support | .477 | .833 | .069 | .572 | .569 | -1.182 | 2.135 |
| | Dentist rated lower denture esthetics | -2.070 | .860 | 245 | -2.408 | .018 | -3.780 | 359 |
| | Perceived pain due to lower denture | .711 | .299 | .253 | 2.374 | .020 | .115 | 1.306 |
| | Patient satisfaction with lower denture retention at rest | 213 | .473 | 064 | 451 | .653 | -1.154 | .727 |
| | Patient satisfaction with lower denture retention at function | 281 | .400 | 115 | 704 | .484 | -1.077 | .514 |
| | Patient satisfaction with lower denture Comfort | .090 | .522 | .033 | .173 | .863 | 948 | 1.128 |
| | Patient satisfaction with easiness of lower denture insertion | 359 | .473 | 068 | 758 | .450 | -1.300 | .583 |
| | Patient general satisfaction with upper and lower dentures | 244 | .518 | 066 | 471 | .639 | -1.275 | .787 |
| | Patient satisfaction with retention of upper and lower dentures during eating | 207 | .504 | 061 | 411 | .682 | -1.211 | .796 |
| | Patient satisfaction with smile<br>and appearance of upper and<br>lower dentures | -1.720 | .888 | 188 | -1.937 | .056 | -3.488 | .047 |
| | Patient satisfaction with retention of upper and lower dentures during speaking | 653 | .366 | 177 | -1.787 | .078 | -1.381 | .074 |

R<sup>2</sup>= Coefficient of determination, DW= Durbin Watson statistic, Unst Co= Unstandardized coefficient, St Co= Standardized coefficient, B= Beta statistics, SE= Standard Error, t= t statistics, P= Two tailed probability value, CI= Confidence intervals. \*Gender, age, having the lower denture carved or not, and dentist ratings of lower dentures, and patient satisfaction with dentures were entered in the regression model.

**Table 7.** Linear regression analyses to predict patient satisfaction with different denture aspects utilizing the demographic variables, having the lower denture carved or not, and dentist ratings of lower dentures among the study sample (n= 50).

| | | Unst | Co | St Co | | | 95% C | I for B |
|---|---|---|---|---|---|---|---|---|
| Dependent | | | | | | | Lower | Upper |
| variable | Predictors* | В | SE | Beta | t | P | Bound | Bound |
| Patient | Constant | 6.768 | 3.155 | | 2.145 | .035 | .499 | 13.038 |
| satisfaction | Gender | .970 | .449 | .222 | 2.163 | .033 | .079 | 1.862 |
| with lower | Age | 058 | .026 | 211 | -2.242 | .027 | 109 | 007 |
| denture | Carved denture or not | .338 | .395 | .078 | .856 | .394 | 447 | 1.124 |
| retention at | Dentist rated lower denture | 170 | .164 | 151 | -1.035 | .303 | 495 | .156 |
| rest | retention | | | | | | | |
| $R^2$ = .295<br>DW=2.000 | Dentist rated lower denture stability | .527 | .249 | .373 | 2.114 | .037 | .032 | 1.022 |
| | Dentist rated lower denture support | .080 | .264 | .038 | .301 | .764 | 446 | .605 |
| | Dentist rated lower denture esthetics | 021 | .273 | 008 | 075 | .940 | 564 | .523 |
| | Perceived pain due to lower denture | 184 | .084 | 216 | -2.184 | .032 | 351 | 017 |
| Patient | Constant | 4.512 | 4.410 | | 1.023 | .309 | -4.249 | 13.273 |
| satisfaction | Gender | 1.404 | .624 | .238 | 2.251 | .027 | .165 | 2.643 |
| with lower | Age | 031 | .036 | 084 | 864 | .390 | 103 | .041 |
| denture | Carved denture or not | 1.144 | .549 | .195 | 2.085 | .040 | .054 | 2.235 |
| retention at | Dentist rated lower denture | 266 | .229 | 175 | -1.158 | .250 | 722 | .190 |
| function | retention | | | | | | | |
| $R^2 = .309$<br>DW=1.728 | Dentist rated lower denture stability | .958 | .335 | .504 | 2.858 | .005 | .292 | 1.623 |
| | Dentist rated lower denture support | 166 | .371 | 059 | 446 | .657 | 904 | .572 |
| | Dentist rated lower denture esthetics | 431 | .382 | 125 | -1.128 | .262 | -1.189 | .328 |
| | Perceived pain due to lower denture | 365 | .112 | 319 | -3.251 | .002 | 588 | 142 |
| Patient | Constant | 6.926 | 3.523 | | 1.966 | .052 | 075 | 13.927 |
| satisfaction | Gender | 1.374 | .501 | .261 | 2.743 | .007 | .378 | 2.369 |
| with lower | Age | 037 | .029 | 112 | -1.290 | .200 | 094 | .020 |
| denture | Carved denture or not | .412 | .441 | .079 | .934 | .353 | 465 | 1.289 |
| Comfort $R^2$ = .394 | Dentist rated lower denture retention | 275 | .183 | 203 | -1.502 | .137 | 638 | .089 |
| DW=2.100 | Dentist rated lower denture stability | .723 | .278 | .426 | 2.600 | .011 | .171 | 1.276 |
| | Dentist rated lower denture support | 345 | .295 | 137 | -1.168 | .246 | 931 | .242 |

| Patient satisfaction with order denture retention Patient satisfaction with pwer and lower denture esthetics Patient general satisfaction with with pper and lower denture esthetics Patient satisfaction with with with retention of patient satisfaction with with per and lower denture denture esthetics Patient satisfaction with with retention of patient satisfaction with pper and lower denture of patient satisfaction with patient satisfaction with patient satisfaction with pper and lower denture satisfaction with pretention of patient satisfaction with pper and lower denture satisfaction of pper and lower denture satisfaction with pper and lower denture satisfaction power denture satisfaction per and lower denture satisfaction power denture satisfaction power denture satisfaction per and lower denture satisfaction power denture satisfacti | | Dentist rated lower denture esthetics | .032 | .305 | .010 | .104 | .917 | 575 | .639 |
|---|---|---|---|---|---|---|---|---|---|
| Satisfaction with each easiness of lower easiness of lower denture entention Dentist rated lower denture esthetics Perceived pain due to lower dentures and lower entention Dentist rated lower denture retention Dentist rated lower denture esthetics Perceived pain due to lower dentures and lower entention Dentist rated lower denture retention Dentist rated lower denture esthetics Perceived pain due to lower denture and lower dentures and lower denture retention Dentist rated lower denture esthetics De | | 1 | 440 | .094 | 430 | -4.682 | <.001 | 626 | 253 |
| with easiness of lower denture chemistrian and perity and lower denture astisfaction with upper and lower denture and lower denture and lower denture astisfaction bentist rated lower denture astisfaction with upper and lower denture astisfaction bentist rated lo | Patient | Constant | 10.809 | 2.225 | | 4.858 | <.001 | 6.388 | 15.229 |
| Carved denture or not 1.072 1.279 1.026 1.265 1.265 1.281 1.28 | satisfaction | Gender | .498 | .316 | .181 | 1.574 | .119 | 130 | 1.126 |
| Dentist rated lower denture retention Dentist rated lower denture retention Dentist rated lower denture stability Dentist rated lower denture 198 1.16 .222 1.125 .264 -1.51 .547 | | | 011 | .018 | 065 | 619 | .538 | 047 | .025 |
| denture retention netention netent | | Carved denture or not | 072 | .279 | 026 | 259 | .796 | 626 | .481 |
| Dentist rated lower denture support Dentist rated lower denture stability Dentist rated lower denture stability Dentist rated lower denture satisfaction with upper and lower denture satisfaction with retention of upper and lower denture support Dentist rated lower denture satisfaction with upper and lower denture satisfaction with upper and lower denture satisfaction with upper and lower denture satisfaction with upper and lower denture satisfaction with upper and lower denture satisfaction on pper and lower denture satisfaction on the content of upper and lower denture satisfaction with upper and lower denture satisfaction with upper and lower denture satisfaction with upper and lower denture satisfaction on the content of upper and lower denture satisfaction with upper and lower denture satisfaction with upper and lower denture satisfaction upper and lower denture satisfaction with upper and lower denture satisfaction with upper and lower denture satisfaction upper and lower denture satisfaction upper and lower denture satisfaction with upper and lower denture satisfaction upper and lower den | | Dentist rated lower denture | 146 | .115 | 206 | -1.265 | .209 | 376 | .083 |
| R2=.121 | | | | | | | | | |
| Dentist rated lower denture esthetics Support Dentist rated lower denture esthetics Perceived pain due to lower 094 095 176 -1.589 .116 212 .024 | $R^2 = .121$ | | .198 | .176 | .222 | 1.125 | .264 | 151 | .547 |
| Dentist rated lower denture esthetics Perceived pain due to lower denture denture general satisfaction with upper and lower denture retention Dentist rated lower denture support | DW=1.973 | Dentist rated lower denture | 393 | .186 | 297 | -2.109 | .038 | 764 | 023 |
| Patient general satisfaction with upper and lower denture Dentist rated lower denture Stability Dentist rated lower denture Stability Dentist rated lower denture esthetics Perceived pain due to lower denture esthetics Stability Dentist rated lower denture esthetics Stability Dentist rated lower denture stability Dentist rated lower denture stability Dentist rated lower denture esthetics Dentist rated lower denture esthetics Stability Dentist rated lower denture esthetics Stability | | support | | | | | | | |
| Patient general satisfaction with upper and lower denture Patient satisfaction with upper satisfaction with upper and lower denture esthetics Patient satisfaction with upper and lower denture satisfaction with upper and lower denture satisfaction Dentist rated lower denture esthetics Dentist rated lower denture esthetics Dentist rated lower denture satisfaction Dentist rated lower denture esthetics Dentist rated lower denture | | Dentist rated lower denture | .263 | .193 | .164 | 1.365 | .176 | 120 | .646 |
| Patient general satisfaction with upper and lower denture satisfaction with tretention of upper and lower dentures and lower dentures attributes attributes attributes attributes attributes and lower denture satisfaction with upper and lower denture and lower denture and lower denture stability Patient satisfaction with upper and lower denture satisfaction with upper and lower denture satisfaction with pretention of upper and lower dentures during eating R²= .223 DW=1.917 Dentist rated lower denture stability Dentist rated lower denture attributes Denti | | | | | | | | | |
| Patient general satisfaction with upper and lower denture and lower dentures are support | | Perceived pain due to lower | 094 | .059 | 176 | -1.589 | .116 | 212 | .024 |
| Gender | | denture | | | | | | | |
| Age | Patient | Constant | 7.778 | 2.976 | | | .011 | 1.865 | 13.692 |
| with upper and lower dentures R²= .228 DW=2.247 Patient satisfaction with eretention of upper and lower dentures atling eating R²= .223 DW=1.917 Patient satisfaction with retention of upper and lower dentures during eating R²= .223 DW=1.917 Patient stated lower denture or not lower denture denture dentures at support Dentist rated lower denture lower denture lower denture eather lower denture lower lower lower denture lower lo | | Gender | 1.361 | .423 | .346 | 3.216 | .002 | .520 | 2.201 |
| Dentist rated lower denture retention Dentist rated lower denture retention Dentist rated lower denture retention Dentist rated lower denture rated lower denture retention Dentist rated lower denture rated lower dent | | | 018 | .024 | 075 | 759 | .450 | 067 | .030 |
| Dentist rated lower denture Stability Dentist rated lower denture Stability Dentist rated lower denture Stability Dentist rated lower denture Stability Stability Dentist rated lower denture Stability Stability Dentist rated lower denture Stability Stability Dentist rated lower denture Stability Stability Dentist rated lower denture Stability Stability Stability Dentist rated lower denture Stability | | Carved denture or not | .323 | .373 | .082 | .867 | .388 | 417 | 1.064 |
| R <sup>2</sup> = .228 Dentist rated lower denture stability Dentist rated lower denture stability Dentist rated lower denture eithetics Dentist rated lower denture esthetics Perceived pain due to lower denture denture .107 .258 .047 .415 .679 .405 .620 .620 | | Dentist rated lower denture | 261 | .154 | 258 | -1.693 | .094 | 568 | .045 |
| DW=2.247 Stability Dentist rated lower denture -1.33 .249 070 533 .596 628 .363 support Dentist rated lower denture .107 .258 .047 .415 .679 405 .620 esthetics Perceived pain due to lower 254 .079 332 -3.207 .002 412 097 denture Constant 8.189 3.235 2.531 .013 1.761 14.617 Satisfaction with retention of upper and lower denture dentures during eating R²= .223 DW=1.917 Dentist rated lower denture .101 .255 .074 .397 .693 406 .609 .609 .608 .7427 .650 .348 .766 .766 | | retention | | | | | | | |
| Dentist rated lower denture support Dentist rated lower denture esthetics Perceived pain due to lower denture satisfaction with retention of upper and lower dentures during eating R²= .223 DW=1.917 Dentist rated lower denture support Dentist rated lower denture .101 .252 .249 .070 .258 .047 .415 .679 .405 .620 .620 | | Dentist rated lower denture | .216 | .235 | .170 | .919 | .361 | 251 | .683 |
| Support Dentist rated lower denture esthetics Perceived pain due to lower denture denture .107 .258 .047 .415 .679 .405 .620 .002 .002 .412 .097 .002 .412 .097 .002 .002 .412 .097 .003 .003 .003 .004 .004 .005 .0 | DW=2.247 | | | | | | | | |
| Dentist rated lower denture esthetics | | Dentist rated lower denture | 133 | .249 | 070 | 533 | .596 | 628 | .363 |
| Patient satisfaction with retention of upper and lower dentures during eating R <sup>2</sup> = .223 DW=1.917 Dentist rated lower denture Dentist rated lower denture Dentist rated lower denture Dentist rated lower denture Constant S.189 S.235 S.235 | | | | | | | | | |
| Perceived pain due to lower denture | | | .107 | .258 | .047 | .415 | .679 | 405 | .620 |
| Patient Constant S.189 3.235 2.531 .013 1.761 14.617 satisfaction with retention of upper and lower dentures during eating R <sup>2</sup> = .223 DW=1.917 Dentist rated lower denture Constant S.189 3.235 2.531 .013 1.761 14.617 S.189 3.246 .229 2.126 .036 .064 1.891 Age | | | | | | | | | |
| Patient satisfaction with retention of upper and lower dentures during eating R²= .223 DW=1.917 Constant 8.189 3.235 2.531 .013 1.761 14.617 Patient satisfaction with satisfaction with with retention of upper and lower denture or not upper and lower denture dentures during eating R²= .223 Age 013 .026 047 477 .634 065 .040 Dentist rated lower denture eating R²= .223 Dentist rated lower denture esthetics 1.101 .255 .074 .397 .693 406 .609 Dentist rated lower denture esthetics 209 .280 084 745 .458 766 .348 | | Perceived pain due to lower | 254 | .079 | 332 | -3.207 | .002 | 412 | 097 |
| Satisfaction with with retention of upper and lower dentures during eating R²= .223 DW=1.917 Gender .978 .460 .229 2.126 .036 .064 1.891 .026 047 477 .634 065 .040 .026 047 477 .634 065 .040 .027 .121 .265 351 1.259 .028 151 987 .326 499 .168 .029 .168 151 987 .326 499 .168 .029 .280 .074 .397 .693 406 .609 .084 427 .650 .650 .650 .650 .650 | | | | | | | | | |
| with retention of upper and lower dentures during eating R <sup>2</sup> = .223 DW=1.917 Age | | | | | | | | | |
| retention of upper and lower dentures dentures eating R <sup>2</sup> = .223 DW=1.917 Carved denture or not .454 .405 .107 1.121 .265351 1.259 Dentist rated lower denture .101 .255 .074 .397 .693406 .609 Stability .255 .074 .397 .693406 .609 Dentist rated lower denture .111 .271 .054 .410 .683427 .650 Dentist rated lower denture .209 .280084745 .458766 .348 | | | | | | | | | |
| upper and lower dentures dentures at lower green tion Dentist rated lower denture retention 166 .168 151 987 .326 499 .168 Dentist rated lower denture during eating R²= .223 Dentist rated lower denture support .101 .255 .074 .397 .693 406 .609 Dentist rated lower denture support .111 .271 .054 .410 .683 427 .650 Dentist rated lower denture esthetics 209 .280 084 745 .458 766 .348 | | Č | | | | | | | |
| Tetention Dentist rated lower denture Comparison of the comparison of the comp | | | | | | | | | |
| | | | 166 | .168 | 151 | 987 | .326 | 499 | .168 |
| during eating R <sup>2</sup> = .223 Dentist rated lower denture $0.111$ .271 .054 .410 .683427 .650 Support Dentist rated lower denture $0.121$ .271 .084745 .458766 .348 | | | | | | | | | |
| eating $R^2$ = .223 Dentist rated lower denture .111 .271 .054 .410 .683 427 .650 .280 .745 .458 766 .348 .480 .348 | | | .101 | .255 | .074 | .397 | .693 | 406 | .609 |
| R <sup>2</sup> = .223 support support | _ | 2 | 111 | 271 | 054 | 410 | 600 | 407 | 650 |
| DW=1.917 Dentist rated lower denture esthetics209 .280084745 .458766 .348 | | | .111 | .2/1 | .054 | .410 | .683 | 427 | .650 |
| esthetics 200 1.004 1.745 1.456 1.760 1.546 | | | - 200 | 280 | - 084 | - 7/15 | 158 | - 766 | 3/18 |
| | | | 20) | .200 | UU <del>1</del> | / <del>-</del> J | . <del>.</del> | /00 | .J <del>.</del> U |
| | | | 320 | .086 | 386 | -3.713 | <.001 | 491 | 149 |

| | denture | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Patient satisfaction with smile and appearance of upper and lower dentures R <sup>2</sup> = .092 DW=1.959 | Constant | 9.960 | 1.298 | | 7.676 | <.001 | 7.382 | 12.539 |
| | Gender | .235 | .184 | .149 | 1.275 | .206 | 131 | .602 |
| | Age | 009 | .011 | 091 | 856 | .394 | 030 | .012 |
| | Carved denture or not | .014 | .163 | .009 | .088 | .930 | 309 | .337 |
| | Dentist rated lower denture retention | 085 | .067 | 209 | -1.264 | .210 | 219 | .049 |
| | Dentist rated lower denture stability | .078 | .102 | .153 | .761 | .449 | 126 | .282 |
| | Dentist rated lower denture support | 112 | .109 | 147 | -1.027 | .307 | 328 | .104 |
| | Dentist rated lower denture esthetics | .115 | .112 | .124 | 1.021 | .310 | 109 | .338 |
| | Perceived pain due to lower denture | 067 | .035 | 219 | -1.952 | .054 | 136 | .001 |
| Patient satisfaction with retention of upper and lower dentures during speaking R <sup>2</sup> = .185 DW=2.367 | Constant | 12.767 | 3.044 | | 4.194 | <.001 | 6.718 | 18.816 |
| | Gender | .702 | .433 | .179 | 1.623 | .108 | 158 | 1.562 |
| | Age | 019 | .025 | 076 | 754 | .453 | 068 | .031 |
| | Carved denture or not | 280 | .381 | 072 | 735 | .464 | -1.038 | .477 |
| | Dentist rated lower denture retention | 009 | .158 | 009 | 055 | .957 | 323 | .305 |
| | Dentist rated lower denture stability | .254 | .240 | .201 | 1.056 | .294 | 224 | .731 |
| | Dentist rated lower denture support | 074 | .255 | 039 | 290 | .773 | 581 | .433 |
| | Dentist rated lower denture esthetics | 462 | .264 | 202 | -1.752 | .083 | 986 | .062 |
| | Perceived pain due to lower denture | | .081 | 309 | -2.903 | .005 | 397 | 074 |

R<sup>2</sup>= Coefficient of determination, DW= Durbin Watson statistic, Unst Co= Unstandardized coefficient, St Co= Standardized coefficient, B= Beta statistics, SE= Standard Error, t= t statistics, P= Two tailed probability value, CI= Confidence intervals. \*Gender, age, having the lower denture carved or not, and dentist ratings of lower dentures were entered in the regression model.